CLINICAL TRIAL: NCT02752204
Title: Torch: A Phase II Study to Determine the Safety and Efficacy of the Dual mTORC Inhibitor AZD2014 and to Investigate Additional Toxicities in Combination With Rituximab in Relapsed/Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: An Evaluation AZD2014 Alone and in Combination With Rituximab in Relapsed/Refractory Diffuse Large B Cell Lymphoma
Acronym: TORCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Bloodwise (Other); AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-212
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed; Refractory; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma | interventions — vistusertib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 (Other): AZD 2014 oral tablets will be given to patients
  Interventions: Drug: AZD 2014
- Stage 2 (Other): AZD 2014 oral tablets and rituximab infusion will be given to patients
  Interventions: Drug: AZD 2014; Drug: Rituximab

INTERVENTIONS:
Drug: AZD 2014 — AZD2014 125mg BD - 2 days on 5 days off in a 28 day cycle
  Other Names: Vistusertib
Drug: Rituximab — Rituximab 375mg/m2 will be administered intravenously on day 1 of a 28 day cycle for a total of 6 cycles.
  Other Names: Mabthera
  Arms: Stage 2

SUMMARY:
The aim of this clinical trial is to see if the drug called AZD2014 is effective and safe to use to treat patients with relapsed or refractory Diffuse Large BCell Lymphoma (DLBCL). The trial will also be looking at combining the antibody (Rituximab) with the drug AZD2014 in a small number of patients to see if this can be done without increasing the toxicity. 36 patients will be recruited to the trial. 30 will receive AZD2014 alone and the remaining 6 will receive AZD2014 plus rituximab. AZD2014 will be given as a 125mg tablet that is to be taken twice a day for 2 days out of every 7 (i.e. on days 1 and 2 of every week). Rituximab will be given via IV infusion on day 1 of every 28 days (once every 4 weeks) for a maximum of 6 cycles.

DETAILED DESCRIPTION:
This is a prospective, single arm, multicentre, phase II clinical trial utilising a two stage design. Stage one will assess the safety and activity of AZD2014 as a single agent in the treatment of DLBCL in 30 patients. Stage two will assess the additional toxicity of combining AZD2014 with Rituximab in an additional 6 patients.

Stage two will be recruited following the full recruitment of stage 1. Stage 2 recruitment will be staggered with 3 patients recruited and their safety data evaluated prior to the recruitment of the remaining 3 patients.

Post treatment biopsies will be requested at relapse in patients receiving rituximab to assess for evidence of synergy.

Once registered to the study, patients will receive AZD2014 125mg bd on an intermittent schedule of 2 days of treatment followed by 5 days with no treatment. Treatment would be on days 1, 2, 8, 9, 15, 16, 22 and 23 of each course 28 days in duration. Treatment is on-going until progression or withdrawal due to toxicity or patient's choice. For the second stage of the trial, rituximab 375mg/m2 will also be administered intravenously on day 1 of the 28 day cycle for a total of 6 cycles in combination with AZD2014.

All patients will be followed for a minimum of 1 year up until disease progression or death.

For patients still on AZD2014 treatment after 1 year (no progression) treatment should still be reviewed at least 3 monthly. Safety, progression and survival data will be collected every 3 months. Assessments should be as per local practice with a CT scan conducted every 3/4 months.

At progression, patients will then be followed up annually for survival data. Tissue, saliva and blood samples will be collected during treatment to determine the activity of AZD2014 on downstream targets, and correlating with response. This will include biopsy tissue from the pre-treatment sample, any biopsy performed on treatment and at relapse post-AZD2014 should this occur

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) relapsing after at least 1 course of potentially curative, anti-CD20 antibody containing regimen (e.g. RCHOP, GCHOP, RGCVP). High grade transformation from low grade lymphoma (e.g. follicular lymphoma, lymphoplasmacytic lymphoma, chronic lymphocytic leukaemia) is permitted. Patients must have relapsed post-ASCT or be considered not suitable for ASCT.
2. Tissue biopsy (or bone marrow trephine if no other tissue available) confirming histology within 3 months of enrolment.
3. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
4. Aged at least 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
6. Females should be using adequate contraceptive measures (as described in the protocol, different for patient receiving rituximab), should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
7. Male patients should be willing to use barrier contraception (i.e. condoms) as described in the protocol, (different for patient receiving rituximab*)
8. Ability to swallow and retain oral medication
9. CT measurable disease with at least 1 lesion having short axis ≥ 1.5cm or splenomegaly ≥ 14cm in cranio-caudal length attributable to relapsed lymphoma
10. Patients must have negative virology for HIV, hepatitis B and hepatitis C prior to trial entry. Patients with an isolated anti-hepatitis B sAg antibody may be entered as this indicates previous vaccination.. These patients MUST have HBV DNA tested.

Exclusion Criteria:

Patients must not enter the study if any of the following exclusion criteria are fulfilled:

1. Prior chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents, and any investigational agents within 14 days of registration (not including palliative radiotherapy at focal sites). Corticosteroids are permitted during screening but should be weaned down to a maximum dose of prednisolone 10mg daily (or equivalent) by day 1 of cycle 1.

   - With the exception of alopecia, any unresolved toxicities from prior chemotherapy should be no greater than CTCAE (Version 4.0) Grade 2 at the time of registration.
2. Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study.
3. Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment.
4. Exposure to potent or moderate inhibitors or inducers of CYP2C8 if taken within the stated washout periods before the first dose of study treatment.
5. Exposure to sensitive or narrow therapeutic range substrates of the drug metabolising enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1), BCRP, OATP1B1, OATP1B3, OCT1 and OCT2 within the appropriate wash-out period (a minimum of 5 x the reported terminal elimination half-life of each drug) before the first dose of study treatment.
6. Previous treatment with any first generation mTORC1 inhibitors (rapamycin, sirolimus, temsirolimus, everolimus) or any dual mTORC1/2 inhibitors (e.g. AZD2014, AZD8055).
7. Patients who have experienced intolerable AEs prejudged by the treating Investigator due to other mTORC1 or mTORC1/2 inhibitors, PI3 kinase inhibitors, or AKT inhibitors.
8. Patients with proven central nervous system (CNS) involvement.
9. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases (e.g., severe hepatic impairment, interstitial lung disease (e.g.bilateral, diffuse, parenchymal lung disease), uncontrolled chronic renal diseases (e.g. glomerulonephritis, nephritic syndrome, Fanconi Syndrome or Renal tubular acidosis) or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, active bleeding diatheses or active infection. Screening for chronic conditions is not required.
10. Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months:

    * coronary artery bypass graft
    * angioplasty
    * vascular stent
    * myocardial infarction
    * angina pectoris
    * congestive heart failure New York Heart Association Grade ≥2
    * ventricular arrhythmias requiring continuous therapy
    * supraventricular arrhythmias including atrial fibrillation, which are uncontrolled
    * haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other central nervous system bleeding
11. Abnormal echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) at baseline (left ventricular ejection fraction [LVEF] <50%).
12. Torsade's de Pointes within 12 months of study entry.
13. Mean (3 consequent ECGs 1 minute apart) resting QTcF and QTcB >470 msec as per local reading.
14. Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age).
15. Patients with Diabetes Type I or uncontrolled Type II (HbA1c >7 mmol/L assessed locally) as judged by the local investigator.
16. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values unless due to underlying NHL infiltration.

    * Absolute neutrophil count <1.5 x 10^9/L (without GCSF / GMCSF support)
    * Platelet count <100 x 10^9/L
    * Haemoglobin <90 g/L (transfusions permissible)
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times the upper limit of normal (ULN) if no demonstrable liver involvement or >5 times ULN in the presence of liver involvement
    * Total bilirubin >1.5 times ULN unless in the presence of Gilbert's syndrome with an elevated indirect fraction
    * Serum creatinine >1.5 times ULN concurrent with creatinine clearance ≤50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times the ULN
17. Current refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD2014.
18. History of known hypersensitivity to active or inactive excipients of AZD2014 or drugs with a similar chemical structure or class to AZD2014.
19. Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
20. Previous history of other active malignant disease other than fully excised basal or squamous cell carcinoma of the skin, carcinoma in situ of the uterine cervix or localised disease treated with curative intent using surgery alone, within the last 3 years.

    For the rituximab cohort only, patients must not enter the study if any of the above or below exclusion criteria are fulfilled:
21. Known hypersensitivity to recombinant proteins, murine proteins or to any excipients of rituximab infusions
22. Vaccination with live virus vaccine within the 4 weeks prior to study entry or intention to do so during the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-07 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Best overall response rate (PR plus CR) (using the Revised Response Criteria for Malignant Lymphoma ) during the first 6 cycles | Data in relation to this outcome will be collected over the first 6 cycles of therapy - each cycle is 28 days in duration

SECONDARY OUTCOMES:
Tolerability rate (based on toxicity assessments using CTCAE v 4.0 criteria) of single agent AZD2014 | Adverse events information will be collected throughout the 18 month recruitment period of the trial and during the one year follow up period
Tolerability rate of additional toxicities when rituximab is combined with AZD2014 at its standard dose (stage 2 only) | Adverse events information will be collected from the start of stage 2 during the 18 month recruitment period of the trial and during the one year follow up period
Best overall response rate post 6 cycles until the end of the trial, assessed using Revised Response Criteria | Information will be collected from cycle 6 ( each cycle is 28 days) during the 18 month recruitment period of the trial until the end of the trial
Overall survival (OS) at 1 year | Information relating to this outcome will be collected up to and including the one year time point
Progression free survival (PFS) at 1 year | Information relating to this outcome will be collected up to and including the one year time point
Duration of response | Information relating to this outcome will be collected throughout the trial during the 18 month recruitment period and during the one year follow up period
Maximum % decrease in the radiological sum of the product of the diameters (SPD) from baseline by CT NCAP | Information relating to this outcome will be collected throughout the 18 month recruitment period of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Graham Collins, MBBS DPhil, Principal Investigator — The Churchill Hospital, Oxford, UK
Locations (9):
- United Kingdom (9):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Liverpool University Hospital, Liverpool
  - University College London Hospitals, London
  - Guys Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich
  - The Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided